CLINICAL TRIAL: NCT05302895
Title: Efficiency of an All-in-one Health Monitoring Device in Elderly Residential Setting
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Haven of Hope Hospital (Other); The Social Innovation and Entrepreneurship Development Fund, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Assistant Professor, The University of Hong Kong
Other Study IDs: HKU_healthmonitor_protocol_v3
Record Dates: First submitted 2022-02-28; First posted 2022-03-31 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Technology
Keywords: Gerontechnology; Smart Healthcare Device; Digital Health Technology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- single-group: The health monitoring data of all the resident participants are measured using traditional device and the all-in-one health monitoring device on the same day for 12 weeks
  Interventions: Device: All-in-one health monitoring device

INTERVENTIONS:
Device: All-in-one health monitoring device — The staff will use the new monitoring device to carry out the health monitoring on every day during the 12-week period. After each round of health monitoring by the traditional and the new devices, the staff will need to fill in log sheets designed by HKU to document the time consumed for the entire process.

SUMMARY:
The study explores the benefits from the application of an all-in-one health monitoring device by care staff in old-age home setting: whether the average time consumed for measuring vital signs (including temperature, blood pressure and SpO2) will be shortened after the adoption of the new device. The study also assesses the satisfaction and perceived usability of the stakeholders towards the all-in-one health monitoring device.

DETAILED DESCRIPTION:
Study design

This is a single-group experimental 10-week trial of comparing the time consumed for measuring health indicators by using the new all-in-one health monitoring device and using the traditional devices, using days as the analysis unit (i.e. comparing the time consumed in two measurements on same days). Before the trial, there will be a 2-week period of device piloting and calibration, so all residents will be measured by the new device for 12 weeks. Views and comments from the operation staff on the usage of the device will also be collected.

Subjects

Care staff and residents in Haven of Hope Woo Ping Care & Attention Home & Haven of Hope Nursing Home will be recruited for the main analysis. If residents are competent in giving consent, both residents and their guarantor, who are responsible for making decisions and signing documents for the residents, will be approached for consent. In cases residents are not competent in giving consents, only their guarantor will be approached for consent.

Procedures

System Installation

The system installation includes the set up of Bluetooth connection between the monitoring device and mobile device, network connection of mobile device, set up of mobile app for system dashboard monitoring, data retrieval and printing out. The service unit and the product supplier shall discuss the installation plan.

Operation protocol preparation

A protocol including the dashboard control and related operations will be prepared for the staff.

Pilot run and calibration

The service unit will invite 3-4 eligible residents to participate in the pilot run. During a routine health monitoring session, 1-2 care staff will use the new device to carry out the measurement, and document any issues that influence the operation. The operation protocol will be revised as necessary.

At the same time, the care staff would conduct artificial intelligence (AI) calibration of the all-in-one health monitoring device with the residents. AI calibration involves using a specific wristband to measure the blood pressure of every resident, so that the app of the device can learn and calibrate the measure for every resident. The time spent and problems encountered during calibration will be documented.

Staff training

A few identical training sessions will be delivered to all care staff which will cover test rationale and instructions of using the monitoring device and the dashboard. The training will be recorded for the staff to re-watch it.

Participants' selection

All residents and care staff who operate daily health monitoring on the selected floors/wards in the residential homes will be invited. Residents' height, age and other basic vital health data will be used for calibration of the all-in-one health monitoring device. No other personal information will be recorded. Before the test, the recruitment staff will introduce the study to these participants and their family caregivers.

Implementation

On each day, the care staff will carry out health monitoring (temperature, blood pressure, and SpO2) with traditional devices (i.e. thermometer and blood pressure meter) and the existing workflow protocol on the participating floor, and the data transfer with a tablet manually. Specifically, the care staff need to go out from the nursing station to visit all the residents' rooms for several rounds and carry out the measurements. After each measurement, they immediately input the data in the tablet. On top of that, they (preferably the same staff or same professional level) will go out in separate rounds and use the new monitoring device to carry out the health monitoring again on the participating floor. The staff will need to login each user's account with the smartphone application before each measurement, and log out after each measurement. Each measurement using the new device takes 30 - 60 seconds. As the data integration has been completed, so that no manual data transfer is needed. After each round of health monitoring by the new device or the traditional devices, the staff will need to fill in log sheets designed by the University of Hong Kong (HKU) to document the time consumed for the entire process. HKU will also monitor the quality of how log sheets are filled together with the investigators of Haven of Hope Christian Service (HOHCS). Towards the end of the testing period, the vital signs collected by traditional devices will be passed to HKU research team for comparing the measurements taken by traditional devices and Dyno50. To ensure anonymity, only the numeric identifiers will be included in the dataset for data analysis. The Dyno50 system will remain a closed system and the abovementioned data required for this study will be provided by the two homes upon consent of the residents and guarantors.

In the qualitative sub-study, the unit IC or his/her designated staff in each of the homes will select by convenience at least 2 residents, 2 staff who operate daily health monitoring, and 1 staff who are responsible for the supervision of the health monitoring procedure for the qualitative interview. Also, 0 - 2 caregivers will be interviewed depending on the availability of caregivers who witnessed the daily operation of the all-in-one health monitoring device, as advised by the participating staff. HKU senior research assistant will be responsible for conducting the interviews. Each semi-structured interviews will take around 30 minutes.

Blinding

Participants and group moderators cannot and will not be blinded to the intervention.

Sample size determination

The sample size is estimated by the current number of residents in the two test sites. In the Woo Ping Care & Attention Home, 24 residents and 5 care staff will be included in this study. In the Haven of Hope Nursing Home, 40 residents and 6 care staff will be included.

Data analyses

In the main trial, paired sample t-test will be used to examine the difference in daily operation time between using the new monitoring device and the traditional devices for the 10-week main trial, adjusting for the number of residents measured. Moreover, paired sample t-test will be used to examine the difference in daily operation time between using the new monitoring device and the traditional devices for the 2-week pilot run and calibration and 10-week main trial, adjusting for the number of residents measured.

The qualitative interview content will be transcribed verbatim in Chinese for further analysis. The qualitative interview transcripts will be analyzed using framework analysis to construct a coherent and logical structure from the classification of many opinions and perceptions of the new health monitoring device. The results will then be discussed and consolidated in the panel meetings with the co-investigators.

ELIGIBILITY:
Inclusion Criteria of care staff for main trial:

* are responsible for the supervision of the health monitoring procedure and those who are responsible for the operation of daily health monitoring

Inclusion Criteria of residents for main trial:

* are able to hold the all-in-one health monitoring device with his/her thumbs and index fingers of both hands under the assistance of the staff

Inclusion Criteria of care staff for qualitative interviews:

* Having participated in the main trial

Inclusion Criteria of residents for qualitative interviews:

* Having participated in the main trial
* Able to verbally communicate in Cantonese as perceived by the staff of the related home

Inclusion Criteria of family members for qualitative interviews:

* Having witnessed the daily operation of the all-in-one health monitoring device

Exclusion Criteria of care staff for main trial:

* None

Exclusion Criteria of residents for main trial:

* Residents with implanted pacemakers and/or implanted cardio-defibrillators (ICDs)

Exclusion Criteria of care staff for qualitative interviews:

* None

Exclusion Criteria of residents for qualitative interviews:

* None

Exclusion Criteria of family members for qualitative interviews:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study populations are residents in Haven of Hope Woo Ping Care & Attention Home, residents in Haven of Hope Nursing Home, and nurses, health workers, and/or family members of the residents
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Average time required for health monitoring operation during the 12-week period | 12 weeks
  The change in average daily operation time from using all-in-one health monitoring device compared to using traditional devices. The daily operation time from using all-in-one health monitoring device is recorded in log sheets by the staff.

SECONDARY OUTCOMES:
Qualitative measure: Perceived acceptance in using all-in-one health monitoring device | at the end of 12-week trial period
  The staff, residents and/or family caregivers answer the following question in a semi-structured qualitative interview:
  1. Was it safe to use the new health monitoring device? (probing: how safe/ unsafe?)
  2. Do you want the new health monitoring device to be bigger or smaller? (probing: What is the problem for the current size? How much bigger/ smaller?)
  3. Was it easy or difficult to use the new health monitoring device? (probing: how easy/ difficult?)
  4. In the first place, to what degree did you expect the service users to comply with using the new health monitoring device?
  5. To what degree did you find the service users to comply with using the new health monitoring device?
Qualitative measure: Perceived benefits in using all-in-one health monitoring device | at the end of 12-week trial period
  The staff, residents and/or family caregivers answer the following question in a semi-structured qualitative interview:
  1. Because of using the new health monitoring device, are there changes in the workflow and manpower logistics of vital signs recording?
  2. Is the workflow of vital signs recording done faster or slower? (probing: how much faster/ slower? if faster, by how much do the time saving meet your expectation?)
  3. Do you find (other) benefits in using the new health monitoring device?
Qualitative measure: Perceived concerns in using all-in-one health monitoring device | at the end of 12-week trial period
  The staff, residents and/or family caregivers answer the following question in a semi-structured qualitative interview:
  1. In the first place, were you concerned about the new health monitoring device?
  2. Did you find these concerns in using the new health monitoring device? (probing: What were the events from which you confirm these concerns? Were the actual concerns larger or smaller than your expectations? If the event was malfunctioning, further probing: how did you or your colleagues fix it? How much time and effort was spent in fixing it?)
  3. Were there any unexpected concerns from using the new health monitoring device? (probing: What were the events from which you discover these concerns?)
  4. What suggestions would you make to future users of this health monitoring device to deal with these concerns?

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Haven of Hope Nursing Home, Hong Kong
  - Haven of Hope Woo Ping Care & Attention Home, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for 10 years.

REFERENCES:
- [Background] Piau A, Campo E, Rumeau P, Vellas B, Nourhashemi F. Aging society and gerontechnology: a solution for an independent living? J Nutr Health Aging. 2014 Jan;18(1):97-112. doi: 10.1007/s12603-013-0356-5. PMID 24402399
- [Background] Carmeli, E. (2009). Aspects of assistive gerontechnology. International Journal on Disability and Human Development, 8(3), 215-218.